CLINICAL TRIAL: NCT06004882
Title: Peripheral Nerve Stimulation of Genicular Nerves Versus Conventional Therapy With Intra-articular Steroid Injection for Chronic Knee Pain: A Prospective, Randomized Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0041; NCI-2023-06513 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Nerve Stimulation; Genicular Nerves; Chronic Knee Pain
MeSH Terms: interventions — Triamcinolone; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (standard steroid injection) (Experimental): Participants will receive 1 standard steroid injection.
  Interventions: Drug: Triamcinolone; Drug: Bupivacaine
- Group 2 (PNS therapy plus 1 standard steroid injection). (Experimental): Participants will receive PNS therapy plus 1 standard steroid injection.
  Interventions: Other: PNS therapy; Drug: Triamcinolone; Drug: Bupivacaine
- Group 3 (PNS therapy plus 1 placebo injection) (Experimental): Participants will receive PNS therapy plus 1 placebo injection.
  Interventions: Other: PNS therapy; Other: Placebo

INTERVENTIONS:
Other: PNS therapy — PNS therapy-NS is a 60-day therapy targeting chronic pain. The procedure involves implanting a small piece of wire next to the nerve causing pain, and the wire is connected to an external device that is then used to apply electric pulses to the nerve, blocking pain signals, for 60 days
  Arms: Group 2 (PNS therapy plus 1 standard steroid injection).; Group 3 (PNS therapy plus 1 placebo injection)
Drug: Triamcinolone — Given by Injection
  Arms: Group 1 (standard steroid injection); Group 2 (PNS therapy plus 1 standard steroid injection).
Drug: Bupivacaine — Given by Injection
  Arms: Group 1 (standard steroid injection); Group 2 (PNS therapy plus 1 standard steroid injection).
Other: Placebo — Given by Injection
  Arms: Group 3 (PNS therapy plus 1 placebo injection)

SUMMARY:
To compare the effects of the following types of therapy on knee range of motion when given to patients with chronic knee pain:

* A standard steroid injection
* Peripheral nerve stimulation (PNS) therapy in combination with a standard steroid injection
* PNS therapy in combination with a placebo injection

Steroid injections are given directly into the knee joints and are considered to be the standard therapy for chronic knee pain. In this study, the injection will be made of the steroid drugs triamcinolone and bupivacaine.

DETAILED DESCRIPTION:
Primary Objectives:

* To compare the mean change in knee range of motion using goniometry from at 30 days (visit 2) from baseline among the three treatment arms.

Secondary Objectives:

* To compare the mean change in knee range of motion using goniometry at 60 days (visit 3) and 90 days (visit 4) from baseline among the three treatment arms.
* To compare changes in knee pain scores (NRS), WOMAC index, use of opioids (measured in morphine milliequivalent), and incidence of complications and adverse effects at 30 days, 60 days, and 90 days from baseline among the three treatment arms

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic knee pain (baseline pain score >=4), seen at Pain Management Center at MD Anderson Cancer Center; if patient has bilateral knee pain, the side with the more severe knee pain will be treated first and counted towards the primary and secondary endpoints
* Patients between ages 18-85 years old
* Patient signed informed consent

Exclusion Criteria:

* Patients with cognitive dysfunction or without capacity to consent
* Patient with recent history (<6 months) of drug or alcohol abuse
* Patients with open skin lesion or undergoing antibiotic therapy for local for systemic infection
* Patients with allergies to local anesthesia, steroids, or adhesives
* Patients who are on opioids for reasons other than knee pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 4.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Saba Javed, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org